CLINICAL TRIAL: NCT05797987
Title: Negative Estrogen Receptor (ER) Expression Assessed by 18F-fluoroestradiol Positron Emission Tomography/Computed Tomography (18F-FES PET/CT) in the Metastatic Breast Cancer (MBC) With ER-positive Primary Tumor
Brief Title: Negative ER Expression Assessed by 18F-FES PET/CT in the MBC With ER-positive Primary Tumor
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-25
Record Dates: First submitted 2023-03-22; First posted 2023-04-04 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- FES negative in MBC: Patients who did not present with any ER-positive lesions were characterized as with negative ER expression in the metastatic stage

SUMMARY:
To investigate the treatment pattern and efficacy of patients with positive primary ER lesion but negative ER expression in MBC using a novel convenient way of 18F-fluoroestradiol positron emission tomography/computed tomography (18F-FES PET/CT).

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with breast cancer (according to International Classification of Diseases 10th Revision) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
* MBC patients who underwent 18F-FES PET/CT at the Fudan University Shanghai Cancer Center between 2010 and 2022
* Patients diagnosed with primary ER-positive tumor and who were yet to receive any systemic therapy during the advanced stage

Exclusion Criteria:

* Patients with incomplete medical records and those diagnosed with secondary primary tumors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MBC patients with ER-positive primary tumor who detected negative ER expression in metastatic disease using 18F-FES PET/CT at the Fudan University Shanghai Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 6 weeks

SECONDARY OUTCOMES:
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Biyun Wang, MD, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] You S, Xie Y, Ji M, Liu C, Zhao Y, Gong C, Hu S, Li Y, Yang Z, Wang B. ER status conversion and subsequent treatment: an assessment of negative ER expression detected by 18F-FES PET in metastatic breast cancer patients with ER-positive primary tumors. Ther Adv Med Oncol. 2023 Dec 15;15:17588359231216093. doi: 10.1177/17588359231216093. eCollection 2023. PMID 38107829